CLINICAL TRIAL: NCT01996085
Title: The Usefulness of Non-invasive Assessment of Haemodynamic Profile in the Diagnosis and Treatment of Hypertension
Brief Title: Non-invasive Haemodynamic Assessment in Hypertension
Acronym: FINE-PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Paweł Krzesiński, MD, PhD, Assistant Lecturer in the Department of Cardiology and Internal Diseases, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: WIM-0000000148
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Arterial Hypertension
Keywords: arterial hypertension; hemodynamics; impedance cardiography; hypotensive therapy
MeSH Terms: conditions — Hypertension | interventions — Lisinopril; Telmisartan; Nebivolol; Indapamide; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemodynamic group (Experimental): The treatment choice based on hemodynamic parameters established with ICG method.
  Monotherapy or combined therapy in case of 1/ complex hemodynamic disturbances and/or 2/ office SBP ≥ 160 mm Hg and/or DBP ≥ 100 mmHg and/or 24-h mean SBP ≥ 140 mm Hg and/or 24-h mean DBP ≥ 90 mm Hg
  Interventions: Drug: lisinopril; Drug: Telmisartan; Drug: Nebivolol; Drug: Indapamide/hydrochlorothiazide; Drug: Amlodipine
- Empiric Group (Active Comparator): The treatment choice based on current guidelines (blinded to ICG).
  Monotherapy or combined therapy in case of office SBP ≥ 160 mm Hg and/or DBP ≥ 100 mmHg and/or 24-h mean SBP ≥ 140 mm Hg and/or 24-h mean DBP ≥ 90 mm Hg
  Interventions: Drug: lisinopril; Drug: Telmisartan; Drug: Nebivolol; Drug: Indapamide/hydrochlorothiazide; Drug: Amlodipine

INTERVENTIONS:
Drug: lisinopril — Angiotensin converting enzyme inhibitor recommended in case of:
  1. "hyperconstrictive" profile (SVRI > 2500-2800 dyn•s•cm-5•m2)
  2. "hyperdynamic" profile (CI > 4.2 l/min/m2 and/or HR > 80/min) and office SBP ≥ 160 mm Hg and/or DBP ≥ 100 mmHg and/or 24-h mean SBP ≥ 140 mm Hg and/or 24-h mean DBP ≥ 90 mm Hg (in combination with nebivolol)
  3. "hypervolemic" profile (man - TFC > 34 1/kOhm; women - TFC > 24 1/kOhm) and office SBP ≥ 160 mm Hg and/or DBP ≥ 100 mmHg and/or 24-h mean SBP ≥ 140 mm Hg and/or 24-h mean DBP ≥ 90 mm Hg (in combination with diuretic)
  4. "balanced" profile
  Arms: Hemodynamic group
Drug: Telmisartan — Angiotensin receptor blocker recommended in terms as for lisinopril in case of its intolerance (e.i. cough)
  Arms: Hemodynamic group
Drug: Nebivolol — Beta-blocker recommended in case of:
  1."hyperdynamic" profile (CI > 4.2 l/min/m2 and/or HR > 80/min)
  Arms: Hemodynamic group
Drug: Indapamide/hydrochlorothiazide — 1. "hypervolemic" profile (man - TFC > 34 1/kOhm; women - TFC > 24 1/kOhm)
  2. "hyperconstrictive" profile (SVRI > 2500-2800 dyn•s•cm-5•m2) and office SBP ≥ 160 mm Hg and/or DBP ≥ 100 mmHg and or 24-h mean SBP ≥ 140 mm Hg and/or 24-h mean DBP ≥ 90 mm Hg (in combination with lisinopril/telmisartan)
  Arms: Hemodynamic group
Drug: Amlodipine — 1/ SVRI > 2800 dyn•s•cm-5•m2 (in combination with lisinopril/telmisartan)
  Arms: Hemodynamic group
Drug: lisinopril — Drug choice at the discretion of physician (blinded to ICG)
  Arms: Empiric Group
Drug: Telmisartan — Angiotensin receptor blocker recommended as for lisinopril in case of its intolerance (e.i. cough)
  Arms: Empiric Group
Drug: Nebivolol — Drug choice at the discretion of physician (blinded to ICG)
  Arms: Empiric Group
Drug: Indapamide/hydrochlorothiazide — Drug choice at the discretion of physician (blinded to ICG)
  Arms: Empiric Group
Drug: Amlodipine — Drug choice at the discretion of physician (blinded to ICG)
  Arms: Empiric Group

SUMMARY:
Arterial hypertension (AH) is an important clinical social and economic problem. In the pathogenesis of AH increased BP is a result of complex mechanisms i. e. fluid retention, increased vascular resistance and hyperkinetic heart function. Impedance cardiography (ICG) is a simple and safe, non-invasive method of hemodynamic monitoring which allows simultaneous assessment of i. e. BP, cardiac index, heart rate, the fluid content in the chest and systemic vascular resistance.

The detailed effect of treatment based on ICG has not been evaluated so far in the long-term observation and for other clinically relevant parameters, such as central blood pressure, left ventricular hypertrophy, metabolic disturbances, parameters of antioxidative-oxidative balance and endothelial function. Therefore, the following main objectives of the study were defined:

* Evaluation of usefulness of impedance cardiography in optimizing treatment of patients with hypertension in the area of reduction and control of blood pressure, hemodynamic parameters, biochemical markers and quality of life.
* Evaluation of complex pathophysiological mechanisms associated with hypertension including hemodynamic, anthropometric, psychological and biochemical parameters as well as the effect of antihypertensive treatment on these phenomena.

The study will be randomized (1:1), prospective and controlled in parallel with conventional treatment. The subjects will be divided into groups according to the pre-established random order:

1. empiric group (GE), in which treatment choice will be based on clinical data and current guidelines
2. hemodynamic group (HD), in which treatment choice will be based on clinical data and current guidelines considering hemodynamic parameters established with ICG method.

All patients will undergo a detailed examination three times: before treatment, then after 3 and 12 months of treatment.

The authors expect that the study will consolidate the importance of ICG in the diagnosis of patients with AH. Simultaneous multiparametric evaluation of the subjects guarantees a unique and innovative results which can enhance our knowledge in pathophysiology of AH and reversibility of adverse mechanisms associated with this disease.

DETAILED DESCRIPTION:
THE IMPORTANCE OF THE PROJECT. Arterial Hypertension (AH) is an important clinical social and economic problem and a major risk factor of coronary artery disease, heart failure, kidney failure and stroke. The risk of organ damage can be significantly reduced just by achieving proper control of blood pressure (BP). In the pathogenesis of AH increased BP is a result of complex mechanisms i. e. fluid retention, increased vascular resistance and hyperkinetic heart function. Impedance cardiography (ICG) is a simple and safe, non-invasive method of hemodynamic monitoring which allows simultaneous assessment of i. e. BP, cardiac index, heart rate, the fluid content in the chest and systemic vascular resistance. The studies conducted so far (including the applicant's own studies) have demonstrated that ICG provided a better selection of drugs and their doses in the short-term observation.

The detailed effect of such treatment strategy has not been evaluated so far in the long-term observation and for other clinically relevant parameters, such as central blood pressure, left ventricular hypertrophy, pulse wave velocity, metabolic disturbances, parameters of antioxidative-oxidative balance and endothelial function. Undoubtedly, such an evaluation may be of high importance in evaluating complex pathophysiological mechanisms associated with cardiovascular hemodynamics. It is expected that the results of this study performed in a group representing a large population of hypertensive patients will allow highly objective, multiparametric evaluation of the usefulness of ICG in hypotensive therapy. The conclusions may be clinically, socially and economically important, especially in terms of effectiveness and continuity of treatment in patients with AH and primary prevention of cardiovascular events and organ damage.

THE CONCEPT AND STUDY DESIGN.

The main aims:

1. Evaluation of usefulness of impedance cardiography in optimizing treatment of patients with hypertension in the area of reduction and control of blood pressure, hemodynamic parameters, biochemical markers and quality of life.
2. Evaluation of complex pathophysiological mechanisms associated with hypertension including hemodynamic, anthropometric, psychological and biochemical parameters as well as the effect of antihypertensive treatment on these phenomena.

The specific aims:

1. Evaluation of the added value of the algorithm of treatment based on the ICG in optimizing treatment of patients with AH in the reduction and control of BP, hemodynamic, biochemical markers and quality of life.
2. Optimization of the used algorithm of antihypertensive treatment on the basis of multiparametric clinical evaluation.
3. Determination of hemodynamic profiles of patients with AH including multiparametric clinical evaluation.
4. Evaluation of complex pathophysiological mechanisms associated with AH including hemodynamic, anthropometric, psychological and biochemical parameters.
5. Evaluation of the impact of antihypertensive treatment on the values of the studied haemodynamic and anthropometric parameters, biochemical markers and quality of life.

The study will be randomized (1:1), prospective and controlled in parallel with conventional treatment. Study group will involve 140 patients of both sexes, aged from 18 to 75 years. All patients will undergo a detailed examination three times: before treatment, then after 3 and 12 months of treatment, according to the following protocol.

Qualification visit. Clinical assessment with consideration of the criteria of inclusion and exclusion. Presentation of information on the project.

First visit (after qualification):

* physical examination with particular attention to factors of cardiovascular risk, including BP measurement in accordance with the recommendations,
* standard 12-lead electrocardiogram,
* echocardiography,
* 6-minute walk test (6-MWT),
* impedance cardiography (ICG),
* measurement of central blood pressure by applanation tonometry,
* measurement of ankle-brachial index (ABI),
* ambulatory blood pressure measurement (ABPM),
* assessment of brachial artery vasodilatation after ischemia (FMD),
* laboratory tests [wide range],
* psychological testing,
* anthropometry,
* assessment of hemodynamics of retrobulbar vessels with use of color Doppler imaging (CDI)
* cardiovascular risk assessment - based on the examination and the results of laboratory tests.

At the first visit antihypertensive therapy and non-pharmacological treatment (individualized diet, weight reduction, regular physical activity, ceasing smoking) will be recommended. The subjects will be divided into groups according to the pre-established random order (www.randomization.com):

1. empiric group (GE), in which treatment choice will be based on clinical data and current guidelines;
2. hemodynamic group (HD), in which treatment choice will be based on clinical data and current guidelines considering hemodynamic parameters established with ICG method.

The choice of treatment in GE group will be performed by a research team member blinded to ICG result. The subjects will not be informed about the type of intervention used. The randomization into the study groups - as on the first visit - will be maintained for all visits.

Depending on the values of SVRI, CI, HR and TFC, hemodynamic disturbances are defined as: (1) hemodynamic profile with excessive vasoconstriction (hyperconstrictive, C: in case of SVRI > 2500 dyn•s•cm-5•m2), (2) with hyperdynamic heart function (hyperdynamic, D: CI > 4.2 l/min/m2 and/or HR > 80/min), (3) with characteristics of overhydration (hypervolemic, V: man - TFC > 34 1/kOhm; women - TFC > 24 1/kOhm), (4) balanced hemodynamic profile balanced (B, hemodynamic parameters of thresholds predefined below) - angiotensin converting enzyme inhibitors indicated.

In STEP 1, when the patient's hemodynamic profile will be hyperdynamic - beta-blocker will be recommended, when hypervolemic -diuretic, when hyperconstrictive - angiotensin converting enzyme inhibitor or angiotensin receptor blocker (if systemic vascular resistance index > 2800 dyn•s•cm-5•m2 - angiotensin converting enzyme inhibitor/angiotensin receptor blocker with calcium blocker recommended). In cases of complex hemodynamic disturbances the combined therapy will be applied.

The STEP 2 will be reserved for the patients with relatively high blood pressure (expected reduction ≥ 20/10mmHg, 24-h mean BP ≥ 140/90 mmHg) of when impedance cardiography suggested only one hemodynamic disturbance. They were assumed to demand polytherapy for that reason the second drug will be added to the first chosen in STEP 1 in combinations:

1. beta-blocker with angiotensin converting enzyme inhibitor/angiotensin receptor blocker;
2. angiotensin converting enzyme inhibitor/angiotensin receptor blocker with diuretic;
3. diuretic with angiotensin converting enzyme inhibitor/angiotensin receptor blocker.

Second visit (after 3 months of pharmacotherapy):

* physical examination with particular attention to factors of cardiovascular risk, including BP measurement in accordance with the recommendations,
* impedance cardiography (ICG),
* measurement of central blood pressure by applanation tonometry,
* ambulatory blood pressure measurement (ABPM),
* laboratory tests [narrow range],
* psychological testing,
* anthropometry
* cardiovascular risk assessment - based on the examination and the results of laboratory tests.

Third visit (after 9 months from the second visit, or in cases of hospitalization for cardiovascular reasons): range of examinations and tests as at the first visit, In the course of observation, each patient will have the right to contact research team on his own initiative for questions and concerns related to participation in the study or his health condition.

CHARACTERISTICS OF THE MAIN APPLIED RESEARCH METHODS.

Laboratory tests will be performed at the Department of Laboratory Diagnostics of Military Medical Institute:

1. [wide range]: blood count, ionogram, creatinine, urea, uric acid, alanine aminotranserase and aspartate aminotranserase, creatine kinase (CK, CK-MB), lipid profile: total cholesterol, LDL and HDL cholesterol, triglycerides, fasting glucose, insulin, glycosylated hemoglobin (HbA1C), lipoprotein (a), leptin, adiponectin; urinalysis, microalbuminuria, homocysteine; high sensitive C-reactive protein (hsCRP), coagulogram, fibrinogen, D-dimer, superoxide dismutase, plasminogen activator inhibitor 1, resistin
2. [narrow range]: blood count, ionogram, creatinine, urea, lipid profile, fasting glucose Impedance cardiography (ICG). On the basis of 10-minute rest recordings of ICG the detailed analysis of mean values of hemodynamic parameters will be performed for: systolic blood pressure (SBP), mean blood pressure (MBP), diastolic blood pressure (DBP), pulse pressure (PP), heart rate (HR), stroke volume (SV) and index (SI), cardiac index (CI), systemic vascular resistance index (SVRI), total artery compliance (TAC) and characteristics of aortic flow: velocity index (VI) and acceleration index (ACI).

Final assessment will also include spectral variability of hemodynamic parameters (i. e. HR, CI, SV, SVR).

Central blood pressure measurement (applanation tonometry). Non-invasive assessment of central blood pressure and related parameters will be performed using the method of applanation tonometry (SphygmoCor Px Aortic BP Profile System). The parameters derived from aortic blood pressure waveform analysis such as i.e. aortic augmentation index (AAI), central blood pressure (CBP) and central pulse pressure (CPP) will be analyzed.

Ambulatory blood pressure monitoring (ABPM). All the patients included in the study will undergo ABPM (Spacelabs 90207; Spacelabs, Medical Inc, Redmond, Washington, USA). The average values of SBP, MBP, DBP, PP (derived from 24-h period, daytime and nightime period) and the corresponding standard deviations (SD) will be analyzed. As the minimum acceptable number of valid BP measurements a 70% is assumed.

Echocardiography. Echocardiography will be performed according to current standards with the use of Vivid 7 apparatus (GE-Healthcare, the USA). Measurements connected with size of heart chambers, contractility and left ventricle wall thickness, ejection fraction and left ventricle relaxation disorders will be evaluated and recorded. The examination will also include automated functional imaging (AFI) of left ventricle.

Flow-mediated dilatation (FMD). The measurement will be performed in the morning, in a quiet room after 10 minutes of rest in supine position. Evaluation of the brachial artery will be done in a 2-D projection, 3-5 cm above the cubital fossa, with the Doppler linear probe of frequency 8 MHz. Dilation of the brachial artery after ischemia will be expressed as a percentage change in brachial artery diameter induced by ischemia in relation to the diameter of the vessel prior to ischemia, in accordance with generally accepted methodology.

Color Doppler Imaging (CDI) of retrobulbar vessels and ophthalmic examination Evaluation of the retrobulbar vessels (ophthalmic artery OA, central retinal artery CRA and short posterior ciliary arteries (temporal and nasal) TSPCA, NSPCA) of the randomly selected eye will be done with the Doppler linear probe of frequency 6-15 MHz (LOGIQ 9 Color Doppler Imaging System; General Electric Medical Systems, Milwaukee, Wisconsin, USA) and will include assessment of peak systolic velocity (PSV), end diastolic velocity (EDV) and resistance index (RI) calculated as follows: RI = (PSV -EDV)/PSV.

All subjects underwent also the randomly selected eye examination that included: autorefractometry and air-puff tonometry (TRK-1P, TOPCON Corporation, Tokyo, Japan), slit-lamp and stereo optic disc evaluation and Spectral optical coherence tomography (OCT/SLO) (Ophthalmic Technologies, Inc. OTI, Toronto, ON, CANADA) of the optic nerve head (ONH), retinal nerve fiber layer (RNFL) and macula.

DATA ANALYSIS. All results will be archived in the form of extensive database with the possibility of multiple analysis, using advanced data analysis systems, such as Statistica, SPSS, MedCalc. To evaluate of complex pathophysiological mechanisms associated with hypertension including hemodynamic, anthropometric, psychological and biochemical parameters (well as the effect of antihypertensive treatment on these phenomena) the correlations and inter-subgroups comparisons will be performed. The results of detailed ophthalmic examination will be also referred to cardiovascular assessment.

MEASURABLE DOCUMENTED EFFECT OF THE PROBLEM. The authors expect that the study will form the basis of the substantive merits of implementing the proposed algorithm of hemodynamic assessment in broad clinical practice as a tool supporting optimization of hypotensive therapy. It is expected that the results will consolidate the importance of ICG in the diagnosis of patients with AH. Simultaneous multiparametric evaluation of the subjects guarantees a unique and innovative results which can enhance our knowledge in pathophysiology of AH and reversibility of adverse mechanisms associated with this disease. It may become an inspiration to undertake further clinical trials related to the practical application of new methods of hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* untreated AH (elevated BP values ≥ 3 months) and insufficiently controlled AH by one or two antihypertensive drugs.

Exclusion Criteria:

* confirmed secondary AH,
* improperly controlled AH with three or more medicines
* chronic renal failure in the third and higher stages of the disease,
* other severe concomitant diseases: systolic heart failure, cardiomyopathy, significant cardiac arrhythmia, significant valvular disease, chronic obstructive pulmonary disease (stage C/D), diabetes, previously undetected, polyneuropathy, peripheral vascular disease,
* body mass index (BMI) > 40 kg/m2,
* mental illness, preventing cooperation with the physician,
* heart rhythm other than sinus (including, i.e. constant heart stimulation),

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
24-h mean Systolic Blood Pressure (in ABPM) | after 3 months from recruitment
24-h mean Diastolic Blood Pressure (in ABPM) | after 3 months from recruitment
daytime mean Systolic Blood Pressure (in ABPM) | after 3 months from recruitment
daytime mean Diastolic Blood Pressure (in ABPM) | after 3 months from recruitment
night-time mean Systolic Blood Pressure (in ABPM) | after 3 months from recruitment
night-time mean Diastolic Blood Pressure (in ABPM) | after 3 months from recruitment
Systolic Blood Pressure (in OBPM) | after 3 months from recruitment
Diastolic Blood Pressure (in OBPM) | after 3 months from recruitment
24-h mean Systolic Blood Pressure (in ABPM) | after 12 months from recruitment
24-h mean Diastolic Blood Pressure (in ABPM) | after 12 months from recruitment
daytime mean Systolic Blood Pressure (in ABPM) | after 12 months from recruitment
daytime mean Diastolic Blood Pressure (in ABPM) | after 12 months from recruitment
night-time mean Systolic Blood Pressure (in ABPM) | after 12 months from recruitment
night-time mean Diastolic Blood Pressure (in ABPM) | after 12 months from recruitment
Systolic Blood Pressure (in OBPM) | after 12 months from recruitment
Diastolic Blood Pressure (in OBPM) | after 12 months from recruitment

SECONDARY OUTCOMES:
change from baseline in Systolic Blood Pressure (in OBPM) at 3 months | after 3 months from recruitment
change from baseline in Diastolic Blood Pressure (in OBPM) at 3 months | after 3 months from recruitment
change from baseline in 24-h Systolic Blood Pressure (in ABPM) at 3 months | after 3 months from recruitment
change from baseline in 24-h Diastolic Blood Pressure (in ABPM) at 3 months | after 3 months from recruitment
change from baseline in daytime Systolic Blood Pressure (in ABPM) at 3 months | after 3 months from recruitment
change from baseline in daytime Diastolic Blood Pressure (in ABPM) at 3 months | after 3 months from recruitment
change from baseline in night-time Systolic Blood Pressure (in ABPM) at 3 months | after 3 months from recruitment
change from baseline in night-time Diastolic Blood Pressure (in ABPM) at 3 months | after 3 months from recruitment
change from baseline in Systolic Blood Pressure (in OBPM) at 3 months | after 12 months from recruitment
change from baseline in Diastolic Blood Pressure (in OBPM) at 3 months | after 12 months from recruitment
change from baseline in 24-h Systolic Blood Pressure (in ABPM) at 3 months | after 12 months from recruitment
change from baseline in 24-h Diastolic Blood Pressure (in ABPM) at 3 months | after 12 months from recruitment
change from baseline in daytime Systolic Blood Pressure (in ABPM) at 3 months | after 12 months from recruitment
change from baseline in daytime Diastolic Blood Pressure (in ABPM) at 3 months | after 12 months from recruitment
change from baseline in night-time Systolic Blood Pressure (in ABPM) at 3 months | after 12 months from recruitment
change from baseline in night-time Diastolic Blood Pressure (in ABPM) at 3 months | after 12 months from recruitment

OTHER OUTCOMES:
Heart Rate (HR) | after 3 months from recruitment
Cardiac Index (CI) | after 3 months from recruitment
Thoracic Fluid Content (TFC) | after 3 months from recruitment
Systemic Vascular Resistance Index (SVRI) | after 3 months from recruitment
augmentation index (AAI) | after 3 months from recruitment
Central Systolic Blood Pressure | after 3 months from recruitment
Central Diastolic Blood Pressure | after 3 months from recruitment
Flow-mediated Dilatation (FMD) | after 3 months from recruitment
Heart Rate (HR) | after 12 months from recruitment
Cardiac Index (CI) | after 12 months from recruitment
Thoracic Fluid Content (TFC) | after 12 months from recruitment
Systemic Vascular Resistance Index (SVRI) | after 12 months from recruitment
augmentation index (AAI) | after 12 months from recruitment
Central Systolic Blood Pressure | after 12 months from recruitment
Central Diastolic Blood Pressure | after 12 months from recruitment
Flow-mediated Dilatation (FMD) | after 12 months from recruitment
left ventricular mass index(LVMI) | after 12 months from recruitment
change from baseline in Heart Rate (HR) at 3 months | after 3 months from recruitment
change from baseline in Cardiac Index (CI) at 3 months | after 3 months from recruitment
change from baseline in Thoracic Fluid Content (TFC) at 3 months | after 3 months from recruitment
change from baseline in Systemic Vascular Resistance Index (SVRI) at 3 months | after 3 months from recruitment
change from baseline in augmentation index (AAI) at 3 months | after 3 months from recruitment
change from baseline in Central Systolic Blood Pressure at 3 months | after 3 months from recruitment
change from baseline in Central Diastolic Blood Pressure at 3 months | after 3 months from recruitment
change from baseline in Flow-mediated Dilatation (FMD) at 3 months | after 3 months from recruitment
change from baseline in Heart Rate (HR) at 12 months | after 12 months from recruitment
change from baseline in Cardiac Index (CI) at 12 months | after 12 months from recruitment
change from baseline in Thoracic Fluid Content (TFC) at 12 months | after 12 months from recruitment
change from baseline in Systemic Vascular Resistance Index (SVRI) at 12 months | after 12 months from recruitment
change from baseline in augmentation index (AAI) at 12 months | after 12 months from recruitment
change from baseline in Central Systolic Blood Pressure at 12 months | after 12 months from recruitment
change from baseline in Central Diastolic Blood Pressure at 12 months | after 12 months from recruitment
change from baseline in Flow-mediated Dilatation (FMD) at 12 months | after 12 months from recruitment
change from baseline in left ventricular mass index (LVMI) at 12 months | after 12 months from recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Krzesinski, MD, PhD, Principal Investigator — Department of Cardiology and Internal Diseases, Military Institute of Medicine, Poland
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Background] Ventura HO, Taler SJ, Strobeck JE. Hypertension as a hemodynamic disease: the role of impedance cardiography in diagnostic, prognostic, and therapeutic decision making. Am J Hypertens. 2005 Feb;18(2 Pt 2):26S-43S. doi: 10.1016/j.amjhyper.2004.11.002. PMID 15752931
- [Background] Taler SJ, Textor SC, Augustine JE. Resistant hypertension: comparing hemodynamic management to specialist care. Hypertension. 2002 May;39(5):982-8. doi: 10.1161/01.hyp.0000016176.16042.2f. PMID 12019280
- [Background] Smith RD, Levy P, Ferrario CM; Consideration of Noninvasive Hemodynamic Monitoring to Target Reduction of Blood Pressure Levels Study Group. Value of noninvasive hemodynamics to achieve blood pressure control in hypertensive subjects. Hypertension. 2006 Apr;47(4):771-7. doi: 10.1161/01.HYP.0000209642.11448.e0. Epub 2006 Mar 6. PMID 16520405
- [Background] Ferrario CM, Flack JM, Strobeck JE, Smits G, Peters C. Individualizing hypertension treatment with impedance cardiography: a meta-analysis of published trials. Ther Adv Cardiovasc Dis. 2010 Feb;4(1):5-16. doi: 10.1177/1753944709348236. Epub 2009 Dec 30. PMID 20042450
- [Background] Ferrario CM. New approaches to hypertension management: always reasonable but now necessary. Am J Hypertens. 2005 Feb;18(2 Pt 2):23S-25S. doi: 10.1016/j.amjhyper.2004.11.042. No abstract available. PMID 15752930
- [Background] Krzesinski P, Gielerak G, Kowal J. [Impedance cardiography - a modern tool for monitoring therapy of cardiovascular diseases]. Kardiol Pol. 2009 Jan;67(1):65-71. No abstract available. Polish. PMID 19253194
- [Derived] Krzesinski P, Gielerak G, Stanczyk A, Piotrowicz K, Uzieblo-Zyczkowska B, Banak M, Kurpaska M, Michalczyk L, Jurek A, Wolszczak K, Galas A, Wojcik A, Skrobowski A. The effect of hemodynamically-guided hypotensive therapy in one-year observation: Randomized, prospective and controlled trial (FINEPATH study). Cardiol J. 2016;23(2):132-40. doi: 10.5603/CJ.a2016.0009. Epub 2016 Feb 15. PMID 26876066
- See also: Project's description in national database — http://nauka-polska.pl/dhtml/raporty/praceBadawcze?rtype=opis&objectId=274841&lang=pl